CLINICAL TRIAL: NCT00529412
Title: Bioresorbable Membrane to Reduce Postoperative Small Bowel Obstruction in Patients With Gastric Cancer. A Randomized Clinical Trial
Brief Title: Bioresorbable Membrane to Reduce Postoperative Small Bowel Obstruction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nihon University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NUSM-CC-01
Record Dates: First submitted 2007-09-13; First posted 2007-09-14 (Estimated); Last update posted 2007-09-14 (Estimated); Status verified 2007-06

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Seprafilm

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control (No Intervention): no Seprafilm
  Interventions: Other: Seprafilm
- Seprafilm (Active Comparator)
  Interventions: Other: Seprafilm

INTERVENTIONS:
Other: Seprafilm — two sheets per body

SUMMARY:
To assess whether the use of Seprafilm reduces the rate of small bowel obstruction in patients who underwent surgery for gastric cancer.

DETAILED DESCRIPTION:
Patients with gastric cancer who were scheduled to undergo gastrectomy were randomly assigned to a sodium hyaluronate-based bioresorbable membrane (Seprafilm) group or to a control group. Before closing the abdominal incision, two sheets of Seprafilm membrane were applied to the surface of the small intestine under the middle abdominal wound in the Seprafilm group. The primary end point was the incidence of bowel obstruction. Secondary end points were intraoperative and postoperative morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of gastric cancer
* Operable

Exclusion Criteria:

* Withdrew consent
* Pregnant
* Ascites
* Distant metastasis
* Liver dysfunction (serum total bilirubin >2.0 mg/dL)
* Renal failure (serum creatinine >1.5 mg/dL)
* A past history of small bowel obstruction.

Max Age: 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2003-08; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
incidence of small bowel obstruction | 3 years, more than 6 months after gastrectomy

SECONDARY OUTCOMES:
intraoperative and postoperative morbidity and mortality. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Tadatoshi Takayama, MD, PhD, Study Chair — Department of Digestive Surgery, Nihon University School of Medicine
Locations (1):
- Department of Digestive Surgery, NIhon University School of Medicine, Tokyo, Japan

REFERENCES:
- [Derived] Hayashi S, Takayama T, Masuda H, Kochi M, Ishii Y, Matsuda M, Yamagata M, Fujii M. Bioresorbable membrane to reduce postoperative small bowel obstruction in patients with gastric cancer: a randomized clinical trial. Ann Surg. 2008 May;247(5):766-70. doi: 10.1097/SLA.0b013e3181656d4e. PMID 18438113